CLINICAL TRIAL: NCT00254007
Title: The Serotonin Transporter Gene Polymorphism and Major Depression Following Traumatic Brain Injury
Brief Title: Depression and Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Krista Lanctot, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205-2003
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Depression; Traumatic Brain Injury
Keywords: depression; traumatic brain injury; serotonin transporter; genetic polymorphisms; citalopram
MeSH Terms: conditions — Depression; Brain Injuries, Traumatic | interventions — Citalopram

INTERVENTIONS:
Drug: citalopram (celexa) — 20(1 tablet)-50(2 1/2 tablets) mg/day for a period of 6 or 10 weeks

SUMMARY:
Problem: Depressive symptoms are a common mental health problem following traumatic brain injury (TBI), occurring in up to 87% of patients. Depression following TBI has important consequences including poor functioning, lack of ability to return to work and family activities and prolonged TBI symptoms. The reason depression develops in some patients following TBI is unknown, making treatment difficult.

One type of brain protein that shows genetic differences between people is called the serotonin transporter. People can be divided by whether or not they have a short protein (S allele) or a long protein (L allele) which influences the amount of serotonin transporter. Serotonin is a key brain chemical in depression in many mental/psychiatric illnesses. We think that the genetic differences in the serotonin transporter, that may not make a difference before TBI, may become important after TBI due to the nature of these injuries.

Methods: A consecutive sample of 200 patients attending a TBI clinic who have sustained a mild-to-moderate TBI (American Congress of Rehabilitation Medicine criteria) within the last 2 months will be assessed for the presence of major depression (standard criteria, standardized interview). In phase I, blood samples from patients with mild-to-moderate TBI with depression and without depression will be checked for the presence of the 5-HTTPR genetic difference. This will allow us to study if the S allele is more likely in TBI patients with depression. In phase II, the patients with depression will be treated with the SSRI citalopram for 6 weeks. At 6 weeks, or upon discontinuation of citalopram, depression will be assessed again. This will allow us to study if depressed patients with the S allele respond more poorly to treatment. Persons assessing depression after treatment will not know the genetic makeup of each patient.

Results Expected: If the serotonin transporter genetic difference confers susceptibility to depression following TBI, this will provide important information on what causes depression following TBI and document a risk factor for depression previously unstudied in this population. Also, as SSRI antidepressants are used to treat depression in TBI, this study may identify a subgroup of TBI patients in whom different medications should be given or additional medications are required.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* gender: male or female
* TBI within the last two months
* mild to moderate TBI
* written, informed consent
* depressed group only: diagnosis of major depressive episode using the depression module of the Structured Clinical Interview for the DSM-IV (SCID-IV)

Exclusion Criteria:

* prior TBI or other focal brain disease (stroke, tumor)
* significant acute medical illness, including: drug overdose, severely disturbed liver, kidney, lung, or heart function, anemia, hypothyroidism, uncontrolled diabetes, Parkinson's disease, Huntington's chorea, progressive supranuclear paralysis, brain tumor, subdural hematoma, multiple sclerosis
* a brain CT scan revealing focal lesions that could not be interpreted as consistent with a TBI
* depression group only: contraindications to receiving treatment with citalopram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-07; Primary Completion 2005-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
- Hamilton Depression Rating Scale (HAM-D) | Baseline, 6 weeks and 10 weeks (if applicable)

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI), Rivermead Head Injury Follow-up Questionnaire (RHFQ), General Health Questionnaire (GHQ), Rivermead Post Concussion Disorder Questionnaire (RPDQ) | Baseline, 6 weeks and 10 weeks (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Krista L Lanctot, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Chan F, Lanctot KL, Feinstein A, Herrmann N, Strauss J, Sicard T, Kennedy JL, McCullagh S, Rapoport MJ. The serotonin transporter polymorphisms and major depression following traumatic brain injury. Brain Inj. 2008 Jun;22(6):471-9. doi: 10.1080/02699050802084886. PMID 18465388